CLINICAL TRIAL: NCT01601015
Title: Effectiveness of the Treatment of Tension-type Headache With Manual and Manipulative Therapy in the Perception of Pain and Cervical Motion: a Double-blind, Randomized, Placebo-controlled Clinical Trial.
Brief Title: Effectiveness of the Treatment of Tension-type Headache With Manual and Manipulative Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, PhD, PT, University of Valencia
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: UVT002
Record Dates: First submitted 2012-05-11; First posted 2012-05-17 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Tension-type Headache
Keywords: Tension-type headache, Effectiveness, Manual therapy
MeSH Terms: conditions — Tension-Type Headache | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Manual therapy (Experimental): Manual therapy of Suboccipital soft tissue Inhibition treatment aims to release the suboccipital muscle spasm that maintains the occiput-atlas-axis joint dysfunction.
  Interventions: Other: Manual Therapy
- Occiput-atlas-axis joint manipulation (Experimental): Is bilaterally administered. The aim of restoring the mobility of joints between occiput, atlas and axis, which enables to correct a global joint dysfunction
  Interventions: Other: Manual Therapy
- Combined treatment (Experimental): The group receiving combined treatment received the two previous techniques exactly with the same sequence.
  Interventions: Other: Manual Therapy
- Control group (Placebo Comparator): Control group not receive treatment and stayed in this position for 10 minutes
  Interventions: Other: placebo treatment

INTERVENTIONS:
Other: Manual Therapy — Manual therapy of Suboccipital soft tissue Inhibition is performed with patient in supine position. The patient's head leans against the physiotherapist's hands, which palpate suboccipital muscles by sliding fingertips until contacting posterior arch of atlas. At this point, a deep and progressive gliding pressure is applied, for 10 minutes. The purpose of this technique is to release suboccipital muscle spasm, which can be responsible for the mobility dysfunction of the occiput-atlas-axis joint.
  Other Names: Tension-type Headache
  Arms: Manual therapy
Other: Manual Therapy — Occiput-atlas-axis joint manipulation is performed in the same position as the previous technique. It is bilaterally administered and it consists of 2 phases: firstly, rotation with gentle head decompression with no flexo-extension and slight lateral flexion is performed, followed by small circumductions aimed at increasing arterial viscoelasticity and searching for adequate joint barrier through selective tension; secondly, a high speed thrust manipulation in pure rotation towards the side to be manipulated is performed, with a head helicoidal movement, with the aim of restoring the mobility of joints between occiput, atlas and axis, which enables to correct a global joint dysfunction.
  Other Names: Tension-type Headache; manipulation
  Arms: Occiput-atlas-axis joint manipulation
Other: Manual Therapy — Occiput-atlas-axis joint manipulation is performed in the same position as the previous technique. It is bilaterally administered and it consists of 2 phases: firstly, rotation with gentle head decompression with no flexo-extension and slight lateral flexion is performed, followed by small circumductions aimed at increasing arterial viscoelasticity and searching for adequate joint barrier through selective tension; secondly, a high speed thrust manipulation in pure rotation towards the side to be manipulated is performed, with a head helicoidal movement, with the aim of restoring the mobility of joints between occiput, atlas and axis, which enables to correct a global joint dysfunction.
  Other Names: Tension-type Headache; Manipulation
  Arms: Combined treatment
Other: placebo treatment — The physiotherapist performed the vertebral artery test bilaterally, followed by a two-minute neck massage without lubricants and with no proven therapeutic effect, as a placebo for all study groups.
  The control group received four sessions of placebo treatment, followed by ten minutes of resting position.
  Other Names: Resting position; Tension-type Headache
  Arms: Control group

SUMMARY:
Background. Tension-type headache (TTH) is the most common form of primary headache and it is a real problem for the subjects suffering from it. Until now, physiotherapy treatments have included different techniques combined together, without establishing which of them is more effective.

Objective. The purpose of this study is to know the effectiveness of manipulative and manual therapy treatments, with regard to pain perception and neck mobility in patients with tension-type headache.

Methods: A double-blind, randomized clinical trial was conducted, with 84 patients diagnosed with tension-type headache, divided into three treatment groups -manual therapy, manipulative therapy, and a combination of both techniques-, and a placebo control group. Four treatment sessions were administered during four weeks, with post-treatment assessment, and follow-up at one month. Cervical ranges of motion were assessed (CROM device), as well as pain perception (McGill Pain Questionnaire), and frequency and intensity of headaches (weekly register).

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 65 years
* Diagnosis of frequent ETTH and CTTH
* Having headache episodes on more than 1 day per month
* Headache episodes lasting from 30 minutes to 7 days
* Headaches having at least 2 of the following characteristics:

  * Bilateral location of pain
  * Pressing non pulsating quality
  * Mild or moderate intensity
  * Not aggravated by physical activity
* Sufferers may present photophobia, phonophobia, nausea or vomiting
* Headache may be associated with pericranial tenderness
* Suffering from TTH for over 3 months
* Subjects being under pharmacological control

Exclusion Criteria:

* Patients with infrequent ETTH, and patients with probable TTH in its frequent and infrequent forms.

  * Headache that is aggravated by head movements.
  * Metabolic or musculoskeletal disorders with symptoms similar to headache
  * Previous neck trauma
  * Vertigo, dizziness, arterial hypertension.
  * Joint stiffness, arteriosclerosis or advanced degenerative osteoarthritis
  * Patients with heart devices
  * Patients in process of pharmacological adaptation
  * Excessive emotional tension
  * Neurological disorders
  * Laxity of neck soft tissues
  * Radiological alterations
  * General hypermobility or hyperlaxity
  * Joint instability
  * Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
An individual clinical interview was conducted to collect socio-demographic data and characteristics of headache in a one-month base period (the previous 4 weeks) | up to 4 weeks
  Firstly, socio-demographic data and characteristics of headache were collected during the four weeks prior to the treatment through individual clinical interview carried out by a physiotherapist who did not participate in the outcome assessment nor in the administration of treatments. It included age and sex, location of pain, side dominance of pain, type of pressure, connection with physical activity, frequency, severity of pain, associated symptoms and pain intensity, rated by the patient on the 0-10 Visual Analogue Scale (VAS) (0 = no pain, 10 = most severe pain).

SECONDARY OUTCOMES:
Multidimensional perception of pain, assessed by the McGill Pain Questionnaire | up to 8 weeks
  includes the following aspects: a) sensory, description of pain in time-space terms; b) affective, description of pain in terms of stress, fear and neurovegetative aspects; and c) evaluative, pain described in terms of general assessment. The McGill Pain Questionnaire is validated in Spanish population [13, 14] and it consists of 66 word descriptors divided into 20 groups, including in each group between 2 and 6 adjectives describing pain. Moreover, it includes a section in which patients register the intensity of pain.
Cervical ranges of motion, measured with the CROM-device | up to 8 weeks
  The CROM-device combines a system of inclinometers and magnets set on a head mainframe with a nose-piece (positions like eyeglasses) and it measures angles of flexion, extension, lateral flexion and rotation. As it includes a system of magnets, the CROM must not be used in subjects with heart devices.
Weekly register | up to 7 weeks
  Frequency and intensity of headache, assessed with a seven register weekly. Patients recorded headache frequency as well as intensity of pain measured by the VAS Scale

CONTACTS AND LOCATIONS:
Overall Officials: Gemma Victoria Espí López, PhD, Principal Investigator — Physiotherapy Department. University of Valencia. Spain
Locations (1):
- Gemma V Espí López, Valencia, Valencia, Spain

REFERENCES:
- [Result] Castien RF, van der Windt DA, Grooten A, Dekker J. Effectiveness of manual therapy for chronic tension-type headache: a pragmatic, randomised, clinical trial. Cephalalgia. 2011 Jan;31(2):133-43. doi: 10.1177/0333102410377362. Epub 2010 Jul 20. PMID 20647241